CLINICAL TRIAL: NCT07001475
Title: A Phase Ib, Multicentre, Randomised, Double Blind, Placebo Controlled, 2 Sequence Crossover Trial to Evaluate the Effects of BI 3031185 on Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics in Patients With Borderline Personality Disorder or Attention-deficit/Hyperactivity Disorder
Brief Title: A Study to Test How BI 3031185 is Tolerated by People With Borderline Personality Disorder or Attention-deficit/Hyperactivity Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1516-0003; 2024-514296-17-00 (Registry Identifier: CTIS); U1111-1309-3549 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-06-02; First posted 2025-06-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Borderline Personality Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Borderline Personality Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BPD Sequence 1: BI 3031185 then placebo (Experimental)
  Interventions: Drug: BI 3031185; Drug: Placebo
- BPD Sequence 2: Placebo then BI 3031185 (Experimental)
  Interventions: Drug: BI 3031185; Drug: Placebo
- ADHD Sequence 1: BI 3031185 then placebo (Experimental)
  Interventions: Drug: BI 3031185; Drug: Placebo
- ADHD Sequence 2: Placebo then BI 3031185 (Experimental)
  Interventions: Drug: BI 3031185; Drug: Placebo

INTERVENTIONS:
Drug: BI 3031185 — BI 3031185
Drug: Placebo — Placebo matching BI 3031185

SUMMARY:
This study is open to adults with borderline personality disorder (BPD) and with attention deficit/ hyperactivity disorder (ADHD). The purpose of this study is to find out how a medicine called BI 3031185 is tolerated by people with BPD or ADHD.

Participants with BPD with ADHD are in separate cohorts. Participants from each cohort are put into 2 groups of equal size randomly, which means by chance. Group 1 takes a single dose of BI 3031185 and Group 2 takes placebo. After a 2-week break, Group 1 takes placebo and Group 2 takes a single dose of BI 3031185. Participants take BI 3031185 and placebo as tablets.

Participants are in the study for about 1 to 2 months. They visit the study site 6 times and have 3 phone or video call visits. For 2 of the visits, participants stay overnight at the study site for 2 nights. During all the visits, doctors check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, and non-binary participants, 18 to 45 years of age, both inclusively, at the time of consent
* Meet current Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria as primary diagnosis as assessed by the Mini International Neuropsychiatric Interview (MINI) at screening for borderline personality disorder (BPD) OR attention-deficit/hyperactivity disorder (ADHD)
* Willingness to abstain from alcohol for 24 h, and all other drugs of abuse including cannabis for 72 h prior to Visits 2 and 3 (Day -1). Willingness to abstain from alcohol and cannabis for 72 h after investigational medicinal product (IMP) administration, as well as from all other recreational drugs for the duration of the trial
* Willingness to abstain from prescribed psychostimulants for 72 h prior to Visits 2 and 3 (Day -1) and 24 h following IMP administration Further inclusion criteria apply

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, delusional disorder, autism spectrum disorder, or antisocial personality disorder as confirmed by the MINI
* Any other psychiatric disorder that is not currently stable in symptoms and treatment
* Any substance use disorder within 3 months prior to randomisation (excluding mild alcohol, cannabis, tobacco, and caffeine use disorders); or moderate to severe substance use disorder within the 6 months prior to randomisation (excluding tobacco and caffeine)
* Positive drug screen. Participants with positive cannabis drug tests can be included if they do not meet criteria for moderate or severe cannabis use disorder and the investigator determines that use will not be an impediment to trial participation or accurate data collection
* Concomitant use of psychotropic medication except for the ones below. All other psychotropic medications must be washed out at least 30 days or 5 Half-life time (t1/2) (whichever is longer) before the start of Visit 2 (Day -1)

  1. A single SSRI (selective serotonin re-uptake inhibitor) or SNRI (selective serotonin and norepinephrine re-uptake inhibitor) antidepressant that has been stable in dose and frequency for >3 months prior to randomisation
  2. A single second-generation antipsychotic at a low dose that has been stable in dose and frequency for >3 months prior to randomisation (low dose = 1 thorazine dose equivalent or less, which translates to ≤2 mg/day for risperidone, 5 mg/day for olanzapine, 75 mg/day for quetiapine, 60 mg/day for ziprasidone, and 7.5 mg/day for aripiprazole)
  3. A single sleep medication given as a nightly scheduled medication (not pro re nata) stable in agent and dose for >3 months prior to screening. Allowed sleep medications include: non-benzodiazepine Z sleep medications, antihistamines, melatonin, trazodone, and doxepin
  4. Participants taking psychostimulant medication prescribed as per label for ADHD must stop medication 72 h prior to Visits 2 and 3 (Day -1) and may resume 24 h after receiving the medication dose on the test day (i.e. 5 days total off of prescribed psychostimulant for Visit 2 and 5 days off of prescribed psychostimulant for Visit 3)
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix
* A positive result for any active hepatitis
* Previous randomisation in this trial Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with borderline personality disorder (BPD) reporting adverse events (AEs) deemed by the investigator to be related to the investigational medicinal product (IMP) from IMP administration to End of Study (EoS) | Up to 24 days
Number of participants with attention deficit/hyperactivity disorder (ADHD) reporting AEs deemed by the investigator to be related to the IMP from IMP administration to EoS | Up to 24 days

SECONDARY OUTCOMES:
Number of participants with BPD reporting any AEs from IMP administration to EoS | Up to 24 days
Number of participants with ADHD reporting any AEs from IMP administration to EoS | Up to 24 days

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - Charité Research Organisation GmbH, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universitätsklinikum Jena, Jena
  - Rheinhessen-Fachklinik Mainz, Mainz
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com